CLINICAL TRIAL: NCT00335803
Title: A Comparison Of Subjects With New Daily Persistent Headache (NDPH) And Subjects With Transformed Migraine (TM)
Brief Title: A Research Study To Compare Two Kinds Of Daily Headache
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Other Study IDs: WBY/NDPH-TM/001
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

SUMMARY:
Chronic daily headache has been classified into several categories. One category is of sudden onset and is called New Daily Persistent Headache (NDPH). Another category of daily headache evolves gradually and is called Transformed Migraine (TM). This research study is being conducted to compare people with these two kinds of daily headache in order to improve our understanding of these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 14-65, inclusive
* Diagnosis of NDPH or TM according to the Silberstein-Lipton criteria.
* Ability to read and understand an informed consent form and study procedures

Exclusion Criteria:

* Pregnancy
* Subjects with any disease or condition that would result in unreliable data or confound the data obtained for this study, as determined by the principal investigator.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-03; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: william b young, M.D., Principal Investigator — Jefferson Headache Center
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States